CLINICAL TRIAL: NCT05496907
Title: Developing an Integrated Model of Care for People With Severe Mental Illness and Type 2 Diabetes: the PsychOsis and Diabetes Service Model (PODS)
Brief Title: Psychosis and Type 2 Diabetes Study (PODS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 289799
Record Dates: First submitted 2022-08-02; First posted 2022-08-11 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-08

CONDITIONS: Type 2 Diabetes; Severe Mental Disorder
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): After the participants consent, they will be asked to complete 7 validated questionnaires. An interview will also take place to determine severity of psychiatric symptoms using the Brief Psychiatric Rating Scale. A physical assessment will be conducted including Blood pressure, BMI and Blood Tests for HbA1c, Glucose test, Total Cholesterol, Renal Function.
  Participants in the intervention arm will see the diabetes nurse up to 10 times, during these sessions motivational interviewing will be used to discuss areas to improve, goal setting and action planning. Participants and the nurse will collaboratively discuss practical strategies to improve their HbA1c, blood pressure, cholesterol, BMI and mental health.
  The same measures that were completed at the beginning will be re-assessed again at 6 months.
  Interventions: Behavioral: Diabetes specialist nurse-led collaborative care intervention
- Control (No Intervention): Participants will be asked to complete the same 7 validated questionnaires, the brief psychiatric rating scale and a physical health assessment at the start. The will continue to receive standard care from their usual care professionals. The same measures that were completed at the beginning will be re-assessed again at 6 months.

INTERVENTIONS:
Behavioral: Diabetes specialist nurse-led collaborative care intervention — 10 sessions with a diabetes nurse to help improve physical and mental health outcomes
  Arms: Intervention

SUMMARY:
People with severe mental illness (SMI), defined as psychotic and bipolar disorders, die 17-20 years earlier than the general population, the most common cause of death being cardiovascular diseases (CVD). The major contributor to CVD mortality in SMI is the increased prevalence of type 2 diabetes (T2D) compared to the general population. T2D is a paradigm of a single condition that progresses to multiple conditions. T2D requires annual reviews of 9 diabetes care processes and for patients to adopt multiple self-care tasks to prevent diabetes complications. The 9 diabetes care processes outlined by the NICE guidelines include: 3-6 monthly blood glucose measurement (HbA1c) with targets; blood pressure measurements and targets; annual blood cholesterol measurement; kidney function testing with urinary albumin; kidney function testing with serum creatinine; weight check; smoking status; diabetes annual eye screening; and annual foot examination.

Previous research has focused on upskilling mental health professionals or link workers in diabetes care, however, a primary care led focus to support individuals with T2D and SMI has not been investigated. This is an interventional study in Lambeth south London testing a new model of care for people with SMI and T2D that is led by the community DSN in collaboration with the PN and mental health team within the Hills Brook and Dales Primary Care Network (PCN). StockWELL PCN participants will act as controls. Participants will complete 7 validated questionnaires, a physical examination including a blood test and urine sample and a brief interview either face to face in their GP surgery. The intervention group will be invited to a clinic run by a DSN. Baseline measures will be repeated after 6 months in both groups. An exit interview will be conducted to determine participants thoughts on the intervention. This project has been funded by the Burdett Trust for Nursing.

DETAILED DESCRIPTION:
The research team will approach the potential participants by contacting them directly and sending a invite letter and the participant information sheet to them by post. This contact is in accordance with consent for future contact given as part of a previous study (IRAS: 307600). Local staff resource/direct care team are not involved in the identification or recruitment of participants in this current application. If the participant contacts the research team, an appointment will be made to complete the consent process, this will occur either over the phone or face to face, depending on the participants' preference.

This will be an interventional study with a non-randomised control group of integrated nurse-led intervention with a 6 month follow up. Patients that belong to GP surgeries in the hills, brook and dales PCN, will automatically be put in the intervention arm, whereas patients who belong to a GP in the StockWELL PCN will be placed in the control group. The investigators will aim to recruit 30 participants in each group, so 60 in total.

After the participants consent, they will be asked to complete 7 validated questionnaires (Diabetes Distress Scale, International Physical Activity Questionnaire, Quality of Life Scale, Global Assessment of Functioning, Alcohol Usage Disorders Identification Test, Drug Abuse Screening Test and Empower Up). These can be found in the case report form, and participants answers will be recorded in the case report form. An Interview will also take place to determine severity of psychiatric symptoms using the Brief Psychiatric Rating Scale. This will take place either face to face at the participants GP surgery or over the phone, depending on the participants preference.

A physical assessment will be conducted including Blood pressure (mmHg), BMI (m/kg2), Urinary ACR (mg/mmol), and Blood Tests for HbA1c (mmol/mol), Glucose test (mmol/L), Total Cholesterol (mmol/mol), Renal Function (mL/min), this will be completed at the participants GP surgery by the direct care team.

This information will be written in a case report form and will kept in a locked filling cabinet in James Clerk Maxwell Building, King's College London (KCL). Data from the form will be entered onto the research REDCAP database by the research team.

Intervention group:

Participants from GP practices within the Hills Brooks and Dales PCN will be invited to face to face or virtual clinics with the DSN and PN. During the appointments the DSN and PN will try and help improve the individual's diabetes control by;

* The patients and health professionals will identify specific and measurable goals to work towards, which will be monitored and form part of a care plan.
* Support the patients' self-management for example medication taking.
* Carry out missing care processes or refer the patient to have them done.
* Discuss strategies on how to optimise a healthy lifestyle and how to improve glycaemic control.
* Sign-post patients to activities and support groups that may benefit their mental and physical wellbeing.
* Encourage patients to engage in regular reviews with DSN/PN to monitor progress and to promote proactive treatment amendments.

Control group:

Participants from 5 GPs in the StockWELL PCN will be invited to join the study by the research team. They will receive their usual diabetes and mental health care. If the research team discover any missing care processes, their care team will be made aware.

Follow-up:

The same measures that were completed at the beginning will be re-assessed again at 6 months, these include; 7 validated questionaries (Diabetes Distress Scale, International Physical Activity Questionnaire, Quality of Life Scale, Global Assessment of Functioning, Alcohol Usage Disorders Identification Test, Drug Abuse Screening Test and Empower Up. An Interview will also take place to determine severity of psychiatric symptoms using the Brief Psychiatric Rating Scale. This will take place either face to face at the participants GP surgery or over the phone, depending on the participants preference.

However, the investigators will also include the Patients Global Impression of Change to measure the overall change in quality of life since beginning the study from the patients' perspective.

A physical assessment will be conducted including Blood pressure (mmHg), BMI (m/kg2), Urinary ACR (mg/mmol), and Blood Tests for HbA1c (mmol/mol), Glucose test (mmol/L), Total Cholesterol (mmol/mol), Renal Function (mL/min), this will be completed at the participants GP surgery by the research team.

To evaluate the patients' experience of this new care pathway exit interviews with participants in the intervention group will be conducted by the research team either over the phone or face to face at the participants GP surgery, depending on their preference. This will approximately take 30 minutes. The interviews will be audio recorded and transcribed before being qualitatively analysed by the research team.

If the participant lacks capacity to consent, the investigators will ask them again in a few weeks to see whether capacity has been restored. If the participant still lacks capacity, their clinical team will be asked if there is a potential personal or professional consultee. The research team will contact this person and ask if they are happy to consent on the participants' behalf.

ELIGIBILITY:
Inclusion Criteria:

* All participants will need to have a diagnosis of type 2 diabetes and bipolar affective disorder or psychosis.
* Capacity to consent: if the participant does not currently have capacity to consent, we will ask them again in a few weeks to see whether capacity has been restored. If the participant still lacks capacity, they will be asked to elect a personal consultee nominee to consent on their behalf. If there is not anyone suitable, we will ask their clinical team to nominate a professional consultee. The research team will then contact this person and ask if they are happy to consent on the participants' behalf.
* Participants must be 18 years or older.

Exclusion Criteria

* Adults without an SMI diagnosis.
* Adults with SMI and other types of diabetes, e.g. type 1 diabetes or gestational diabetes (as different management).
* Self-reported pregnancy status (as would require intensive management in a dedicated clinic).
* Dementia.
* Organic psychosis.
* Moderate-severe learning disabilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of Intervention using HbA1c levels | 6 months
  To compare the HbA1c of participants who receive the integrated diabetes nurse-led intervention with a non-randomised control group.

SECONDARY OUTCOMES:
Blood Pressure | 6 months
  The blood pressure of the intervention group will be compared to the control group after six months.
Body Mass Index (BMI) | 6 months
  BMI, which is a person's weight (kg) divided by their height (m) squared (kg/m2), will be compared after 6 months between the intervention and the control group.
Mental Health Outcome | 6 months
  Mental health will be assessed by the brief psychiatric rating scale. This is a seven point scale (1, not present; 2, very mild; 3, mild; 4, moderate; 5, moderately severe; 6, severe; 7, extremely severe). Thus, the range of possible BPRS total scores is from 18 to 126. A higher score would suggest a more severe psychiatrics symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsty Graham, Principal Investigator — King's College London University
Locations (9):
- United Kingdom (9):
  - Herne Hill Group Practice, London
  - Knight's Hill, London
  - Brixton Hill, London
  - Northwood Group Practice, London
  - Binfield Road Practice, London
  - Springfield Medical Centre, London
  - Beckett House, London
  - Grantham Practice, London
  - Stockwell Group Practice, London

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data can be shared if requested.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Once the study is completed.
Access Criteria: Email Kirsty Winkley to request access.